CLINICAL TRIAL: NCT06338033
Title: Prognostic Study of Visceral Fat and Heart Failure With Preserved Ejection Fraction
Status: Completed | Type: Observational
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dongying Zhang, Clinical Professor, Chongqing Medical University
Other Study IDs: 2024-03-23
Record Dates: First submitted 2024-03-23; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2023-04

CONDITIONS: Heart Failure With Preserved Ejection Fraction and Visceral Fat

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- VFA/BMI<5.49
- VFA/BMI≥5.49

SUMMARY:
Obesity and heart failure with preserved ejection fraction (HFpEF) have multiple pathologic associations that affect the prognosis of HFpEF. Chinese people are more prone to visceral obesity, resulting in varying degrees of true obesity in individuals with the same body mass index (BMI). There are no prognostic studies of VFA/BMI in the HFpEF population.

DETAILED DESCRIPTION:
A total of 298 patients with HFpEF who were hospitalized in the Department of Cardiovascular Medicine of the First Affiliated Hospital of Chongqing Medical University from September 2020 to August 2023 were included in this prospective cohort study.All patients were followed up on November 30, 2023.The primary endpoint of the study was all-cause mortality and secondary endpoints were rehospitalization for heart failure and composite endpoints of both.After a median follow-up of 564 days, a total of 30 (10.1%) patients died and 82 (27.5%) were rehospitalized for heart failure. Patients with HFpEF were categorized into two groups according to median VFA/BMI (VFA/BMI <5.49; VFA/BMI ≥5.49).The aim of this study was to elucidate whether VFA/BMI has prognostic value in patients with HFpEF by Kaplan-Meier survival analysis and cox regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adule aged≥18 years old;
* Diagnosed with HFpEF.

Diagnostic criteria including:

1. left ventricular ejection fraction ≥50%;
2. with signs and/or symptoms of heart failure;
3. Sinus rhythm：BNP≥35pg/mL and/or NT-proBNP≥125pg/mL;Atrial fibrillation rhythm：BNP≥105pg/mL and/or NT-proBNP≥365pg/mL；
4. at least one additional criterion: relevant structural heart disease(LVH and/or LAE) or diastolic dysfunction.

Exclusion Criteria:

* Age ≤18 years;
* malignant tumor;
* comorbid severe hepatic and/or renal insufficiency;
* lost to follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure with preserved ejection fraction(HFpEF)
Sampling Method: Non-Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2020-09-19 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | November 30, 2023
  All-cause mortality

SECONDARY OUTCOMES:
Rehospitalization for heart failure | November 30, 2023
  Rehospitalization for heart failure

OTHER OUTCOMES:
Composite endpoints of all-cause mortality and rehospitalization for heart failure | November 30, 2023
  Composite endpoints of all-cause mortality and rehospitalization for heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Dongying Zhang, doctor, Study Director — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: No